CLINICAL TRIAL: NCT02747966
Title: Study of Access Flow ,Access Recirculation of Arteriovenous Fistula and the Relationship With Cardiac Function
Brief Title: The Relationship Between the Flow of Arteriovenous Fistula and Cardiac Function in Haemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xue Qing Yu, Director, Sun Yat-sen University
Other Study IDs: SYSU-HD02
Record Dates: First submitted 2015-05-21; First posted 2016-04-22 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Complication of Hemodialysis
Keywords: access flow; access recirculation; cardiac output; cardiac index; hemodialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A prospective longitudinal surveillance for a period of 2 months. Sample - identify suitable Chronic Kidney Disease (CKD) patients who undergo HD with functioning AVF. Participants at various age range and both sexes are recruited to observe their access flow, access recirculation and cardiac function and assess their relationship.

DETAILED DESCRIPTION:
All patients recruited who met the inclusion criteria were investigated access flow, access recirculation and cardiac function(including cardiac output,cardiac index,central blood volume,et al).Measurement time is the beginning of HD session (first 30min to 1 hr),Middle of HD session (optional),and the end of the HD session (1hr to 30 min prior to end of session). The follow-up duration is 6 months and 12 months.Repeat the assessment at the above time points.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergo HD with native AVF
* AF of AVF between 300ml/min and 1800ml/min

Exclusion Criteria:

* Patients whose AVF developed Access Recirculation (AR) which cannot be resolved at the time of measurement
* Patients developed access or systemic infection during the study period

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All eligible participants are recruited according the inclusion and exclusion criteria.Their basis data are documented and the central hemodynamic condition are assess cross-sectionally and longitudinally.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
to access the chang of the fistula blood flow in HD patients using Ultrasound Dilution method | Change of the fistula blood flow from baseline to 6 months

SECONDARY OUTCOMES:
Changes of the Cardiac Index (CI) during the course of hemodialysis therapy | from baseline to 6 months
Changes of the Oxygen delivery ( Adequacy of hemoglobin level to Epoetin) during the course of hemodialysis therapy | from baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Xueqing Yu, MD, Principal Investigator — Department of Nephrology, 1st Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The 1st Affiliated Hospital, Sun Yet-sen University, Guangzhou, Guangdong, China